CLINICAL TRIAL: NCT00439179
Title: BrUOG-PA-205 A Phase I Trial of GW572016, Gemcitabine and Oxaliplatin for Metastatic Pancreaticobiliary Cancer Schema GSK Study ProtocolGSK #103556
Brief Title: A Trial of GW572016, Gemcitabine and Oxaliplatin for Metastatic Pancreaticobiliary Cancer Schema
Acronym: BrUOG-PA205
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, howard safran, Principal Investigator, Brown University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-PA-205
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — KPNA1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): Weekly gem + GW572016, 1000mg/day (combination)
  Interventions: Drug: cohort 1
- Cohort 2 (Experimental): Weekly gem + GW572016, 1500 mg/day (combination)
  Interventions: Drug: cohort 2
- cohort 3 (Experimental): GEMOX + GW572016 1000 mg/day (combination)
  Interventions: Drug: cohort 3
- cohort 4 (Experimental): GEMOX + GW572016 1500 mg/day (combination)
  Interventions: Drug: cohort 4

INTERVENTIONS:
Drug: cohort 1 — Weekly gem + GW572016, 1000mg/day (combination)
  Arms: Cohort 1
Drug: cohort 2 — Weekly gem + GW572016, 1500 mg/day (combination)
  Arms: Cohort 2
Drug: cohort 3 — GEMOX + GW572016 1000 mg/day (combination)
  Arms: cohort 3
Drug: cohort 4 — GEMOX + GW572016 1500 mg/day (combination)
  Arms: cohort 4

SUMMARY:
A Phase I Trial of GW572016, Gemcitabine and Oxaliplatin for Metastatic Pancreaticobiliary Cancer Schema

DETAILED DESCRIPTION:
The primary objective of this phase I study is to determine the safety, tolerability and optimal tolerated regimen of GW572016 when combined with gemcitabine and with the combination of gemcitabine and oxaliplatin. Three to six patients will be treated at each dose level to assess toxicity. To better assess the safety at the final dose level in both Stage I and Stage II, the number of patients in the cohort at the Maximum Tolerated Dose for both Stages will be expanded to 10. Therefore approximately 34-37 patients will be treated on this study.

Trial finished and no further data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients are required to have histologically or pathologically confirmed, metastatic or locally advanced adenocarcinoma of the pancreas or biliary tree
* No prior systemic chemotherapy for locally advanced or metastatic pancreaticobiliary cancer. No prior EGFR inhibitors.
* ECOG performance status 0-2 retain ability to swallow oral medications
* Age > 18, non pregnant. Because no dosing or adverse event data are currently available on the use of GW572016 in patients <18 years of age, children are excluded from this study.
* The effects of GW572016 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

A female is eligible to enter and participate in the study if she is of:

1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who:

   * Has had a hysterectomy,
   * Has had a bilateral oophorectomy (ovariectomy),
   * Has had a bilateral tubal ligation, or
   * Is post-menopausal(a demonstration of total cessation of menses for ³1 year).
2. Childbearing potential, has a negative serum pregnancy test at screening, and agrees to one of the following:

   * Intrauterine Device (IUD),
   * Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
   * Complete abstinence from sexual intercourse for two weeks before exposure to investigational products, throughout the clinical trial, and for at least one week after the last dose of investigational product.
   * Double barrier contraception (condom with spermicidal jelly, foam, suppository, or film; diaphragm with spermicide; or male condom and diaphragm)

     * Adequate hematologic function: ANC≥1500/ul,platelets≥100,000/ul,hemoglobin 8
     * Adequate hepatic function with total bilirubin ≤ 1.5mg/dL and ALT or AST ≤ 2x ULN. (Patients with liver metastases may have AST/ALT less than or equal to 5x upper limit of normal). Patients with elevated bilirubin secondary to biliary obstruction that have subsequently been stented may enter the protocol with a bilirubin of < 2.0 as long as the bilirubin is falling.
     * Adequate renal function: (creatinine ≤1.5mg/dL or estimated creatinine clearance greater than 60ml/min calculated by the Cockcroft Formula).
     * Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram or MUGA scan. Note that baseline and on treatment scans should be performed using the same modality and preferably at the same institution.
     * No peripheral neuropathy for patients who receive oxaliplatin.
     * Life expectancy of at least 12 weeks
     * Signed informed consent

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Prior treatment with GW572016 or any EGFR targeting therapies.
* Prior treatment with systemic chemotherapy for metastatic pancreaticobiliary cancer.
* Evidence of brain metastases or leptomeningeal disease
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known contraindications to the use of oxaliplatin or gemcitabine.
* History of allergy to platinum compounds in patients receiving oxaliplatin. Amendment #2 4/28/05
* The subject has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with GW572016
* Participation in any investigational study within 28 days prior to study enrolment
* Any major surgery (insertion of a vascular access device is not considered a major surgery), hormonal therapy (other than replacement), chemotherapy or radiotherapy within the last 4 weeks and/or not recovered from prior therapy within the last 4 weeks and/or not recovered from prior therapy.
* Pregnant or lactating females are excluded from this study because GW572016 is member of the 4-anilinoquinazoline class of kinase inhibitors with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with GW572016, breastfeeding should be discontinued if the mother is treated with GW572016.
* Malabsorption syndrome disease significantly affecting gastrointestinal function or major resection of the stomach or small bowel that could affect absorption of GW572016.
* Any unresolved bowel obstruction.
* The patient has inadequate venous access in the clinical judgment of the investigator or designated clinical staff.
* The patient is taking any medication on the prohibited medications list in Section 10.2 Patients requiring oral anticoagulants (coumadin, warfarin) are eligible provided there is increased vigilance with respect to monitoring INR. If medically appropriate and treatment available, the investigator may also consider switching these patients to LMW heparin, where an interaction with GW572016 is not expected.
* Patients may not be receiving any other investigational agents or receiving concurrent anticancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: howard Safran, MD, Principal Investigator — Brown University
Locations (1):
- Brown University Oncology Research Group, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with both pancreatic and bilary cancer were enrolled
Groups:
- Cohort 1: Cohort 1: Weekly gem + GW572016, 1000mg/day. (combination)
- Cohort 2: Cohort 2: Weekly gem + GW572016, 1500 mg/day. (combination)
- Cohort 3: Cohort 3: GEMOX + GW572016 1000 mg/day. (combination)
- Cohort 4: Cohort 4: GEMOX + GW572016 1500 mg/day.(combination)
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 3 (1 with biliary) | 13 (2 with biliary) | 6 (2 with biliary) | 5 (2 with biliry)
Completed | 3 | 11 | 6 | 5
Not Completed | 0 | 2 | 0 | 0
Not completed — * 1 pt inelig, 1 pt numb not used | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: participant number correlates to all enrolled patients treated on this study as a whole which is the way in which the abstract was written and therefore how these results are entered
Groups:
- Cohort 1: Cohort 1: Weekly gem + GW572016, 1000mg/day.
- Cohort 2: Cohort 2: Weekly gem + GW572016, 1500 mg/day.
- Cohort 3: Cohort 3: GEMOX + GW572016 1000 mg/day.
- Cohort 4: Cohort 4: GEMOX + GW572016 1500 mg/day
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 3 | 11 | 6 | 5 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 4 | 3 | 12
  >=65 years | 1 | 8 | 2 | 2 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (17) | 66 (11) | 61.5 (6) | 64.2 (12) | 63.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 3 | 3 | 11
  Male | 2 | 7 | 3 | 2 | 14
Region of Enrollment [Number; unit: participants]
  United States | 3 | 11 | 6 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Toxicity (Number of Patients Who Experiened DLTs)
Description: To determine the safety and tolerability of GW572016 when administered with gemcitabine and the combination of gemcitabine and oxaliplatin in patients with advanced pancreaticobiliary cancers. Numbers below are DLTs
Time Frame: until death, approximately 2 years
Measure: Number; unit: participants
Groups:
- Cohorts 1: Cohort 1: Weekly gem + GW572016, 1000mg/day.
- Cohort 2: weekly gem+ GW572016, 1500mg/day
- Cohort 3: GEMOX+ GW572016 1000mg day
- Cohort 4: GEMOX+ GW572016 1500mg/day
Arm/Group | Cohorts 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 11 | 6 | 5
participants | 0 | 1 | 1 | 2

2. Secondary Outcome: Number of Patients Who Experienced a Partial Response
Description: To assess clinical activity of GW572016 with gemcitabine and with the combination of gemcitabine and oxaliplatin in patients with advanced pancreaticobiliary cancers.
Time Frame: every two months until progression
Measure: Number; unit: participants
Arm/Group | Cohorts 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 11 | 6 | 5
participants | 0 | 2 | 1 | 1

ADVERSE EVENTS:
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/11 | 0/6 | 1/5
Other Adverse Events (participants affected / at risk) | 0/3 | 1/11 | 1/6 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=11) | Cohort 3 (N=6) | Cohort 4 (N=5)
Gr 3 Infection (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Gr 2 Fever, Gr 1 Chills & Hyperbillirubinemia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=11) | Cohort 3 (N=6) | Cohort 4 (N=5)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — DLT
Fatigue (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nausea (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
anorexia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No